CLINICAL TRIAL: NCT01484132
Title: Health Effects of Dental Composites in Children
Brief Title: Composites and Urinary Bisphenol-A Study
Acronym: CUBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01ES019155 (NIH)
Record Dates: First submitted 2011-11-16; First posted 2011-12-02 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-03

CONDITIONS: Dental Caries
Keywords: Dental Caries; Dental Restorative Materials; Dental Composite; Bisphenol-A
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Composite (Experimental)
  Interventions: Procedure: Restoration of dental caries with dental composite

INTERVENTIONS:
Procedure: Restoration of dental caries with dental composite — Dental Restoration (bisphenol A diglycidyl ether methacrylate based composite)
  Other Names: Composite to be used is Z100 by 3M ESPE (St Paul, MN, USA).

SUMMARY:
The Composites and Urinary Bisphenol-A Study (CUBS) is a clinical study of dental composite for its effects on urinary bisphenol-A levels. The study will enroll approximately 139 children recruited from study-affiliated clinical sites in New England.The primary aim of CUBS is to test the hypothesis that urinary bisphenol-A (BPA) concentrations increase after composite restoration placement. BPA is a chemical used in the synthesis of matrix monomers and has been shown to have harmful effects in toxicological studies in laboratory animals. Currently it is unknown whether dental composite restorative materials containing monomers that are derived from BPA result in chronic low-dose BPA exposure in children.

DETAILED DESCRIPTION:
Study subjects will be new or existing patients of the clinical sites who are in need of dental restorations, meet all eligibility criteria, and provide informed consent/assent to participate. Subjects will be asked to provide two pre-treatment urine samples and three post-treatment samples. Urine collections occur next-day and 14 days after treatment, with one final urine collected approximately 6 months later (marking the end of the subject's active study participation). Data will be collected from the clinician's standard oral examination (including new and existing dental treatments), the data collector's measurements of height and weight and interviews administered to the parents/guardians to assess sociodemographic and other relevant factors (e.g., recent food/beverage consumption). Confidentiality will be maintained by assigning each subject a unique number and using only this number or aggregate data in all study reports. All study records will be securely maintained with access limited to essential study personnel only.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-16 (<17) years at enrollment.
* 2+ posterior teeth with caries requiring restorations treatable by composite.
* Toilet-trained (not using diapers, pull-ups, or training pants during day or night).

Exclusion Criteria:

* Medical conditions that would render the subject physically unable to provide urine samples.
* Guardian is not proficient in spoken English or Spanish language
* Child is aged 8.0 years or older and not proficient in spoken English or Spanish language
* Living >35 miles outside of the dental clinic or the NERI office (Watertown MA)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja McKinlay, PhD, Principal Investigator — Carelon Research
Locations (1):
- New England Research Institutes, Inc., Watertown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 113 children aged 3-17 were enrolled in Composites and Urinary Bisphenol-A Study (CUBS) across 8 dental clinics in Massachusetts between February 2012 and December 2013. Follow-up visits were completed in June 2014.
Period: Overall Study
Arm/Group | Composite
Started | 113
Pre-treatment Urine Sample | 101 (Urine samples were collected twice pre-treatment. 101 subjects completed at least one urine sample.)
Completed | 91 (91 subjects had at least one pre-treatment and at least one post-treatment urine sample.)
Not Completed | 22
Not completed — Lost to Follow-up | 8
Not completed — Difficulty with time commitment | 2
Not completed — Ineligible | 1
Not completed — No pre-treatment urine sample collected | 1
Not completed — No post-treatment urine sample collected | 10

BASELINE CHARACTERISTICS:
Population: 98 of 101 subjects who had the pre-treatment urine sample completed the baseline interview. Therefore, 98 subjects were included in the baseline analysis.
Arm/Group | Composite
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.36 (3.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 52
Race/Ethnicity, Customized [Number; unit: participants]
  White - Non Hispanic | 27
  Black - Non Hispanic | 19
  Hispanic | 38
  Other | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Bisphenol A Level (BPA) From Baseline to 6 Months
Description: BPA was measured, corrected for specific gravity, in ng/mL. We corrected BPA for specific gravity (SG) using the formula: BPA * [(meanSG - 1)/(SG - 1)], where meanSG is the mean of the SG for the samples examined. Urine samples were collected twice pre-treatment and the geometric mean of BPA at each pre-treatment visit was used as the baseline BPA. Change in BPA was computed using BPA at follow-up minus BPA at baseline. Analysis of change in BPA was done using the arithmetic mean.
Time Frame: From Baseline to 6 months
Population: Of 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample, 77 subjects who had BPA at 6 months were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Composite
Number analyzed (Participants) | 77
ng/mL | 0.29 (4.66)
Statistical Analysis 1: Comparison: Composite; One sample t-test was used to test whether the mean change from baseline to 6 months was different from 0; Test type: Superiority or Other; p = 0.58, t-test, 2 sided
Statistical Analysis 2: Comparison: Composite; To see the association between composite exposure on all surfaces and change in BPA from baseline to 6 months, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.406, Regression, Linear — P-value is to test the association between composite exposure on all surfaces and change in BPA from baseline to 6 months after adjusting for covariates; Composite exposure on all surfaces was used as the main predictor and baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.061, 95% CI 2-sided [-0.206 to 0.084]
Statistical Analysis 3: Comparison: Composite; To see the longitudinal association between composite exposure on all surfaces and change in BPA from baseline, the repeated measure model was used with all available follow-up BPA data. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.693, Mixed Models Analysis — P-value is to test the longitudinal association between composite exposure on all surfaces and change in BPA after adjusting for covariates; [statistical method as in outcome 1, analysis 2]; Slope = -0.017, 95% CI 2-sided [-0.101 to 0.067]
Statistical Analysis 4: Comparison: Composite; To see the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 6 months, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.160, Regression, Linear — P-value is to test the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 6 months after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.123, 95% CI 2-sided [-0.296 to 0.050]
Statistical Analysis 5: Comparison: Composite; To see the longitudinal association between composite exposure on posterior occlusal surfaces and change in BPA from baseline, the repeated measure model was used with all available follow-up BPA data. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.574, Mixed Models Analysis — P-value is to test the longitudinal association between composite exposure on posterior occlusal surfaces and change in BPA after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.029, 95% CI 2-sided [-0.131 to 0.073]

2. Primary Outcome: Change in Urinary Bisphenol A Level (BPA) From Baseline to 1 Day After the First Dental Treatment
Description: BPA was measured, corrected for specific gravity, in ng/mL. We corrected BPA for specific gravity (SG) using the formula: BPA * [(meanSG - 1)/(SG - 1)], where meanSG is the mean of the SG for the samples examined. Urine samples were collected twice pre-treatment and the geometric mean of BPA at each pre-treatment visit was used as the baseline BPA. Change in BPA was computed using BPA at 1 day after the first dental treatment minus BPA at baseline. The first dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically within a few weeks of baseline. Analysis of change in BPA was done using the arithmetic mean.
Time Frame: From Baseline to 1 day after the first dental treatment (The first dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically within a few weeks of baseline.)
Population: Of 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample, 89 subjects who had BPA at 1 day after the first dental treatment were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Composite
Number analyzed (Participants) | 89
ng/mL | 1.71 (9.94)
Statistical Analysis 1: Comparison: Composite; One sample t-test was used to test whether the mean change from baseline was different from 0; Test type: Superiority or Other; p = 0.11, t-test, 2 sided
Statistical Analysis 2: Comparison: Composite; To see the association between composite exposure on all surfaces and change in BPA from baseline to 1 day after the first treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.003, Regression, Linear — P-value is to test the association between composite exposure on all surfaces and change in BPA from baseline to 1 day after the first treatment after adjusting for covariates; [statistical method as in outcome 1, analysis 2]; Slope = 0.299, 95% CI 2-sided [0.105 to 0.494]
Statistical Analysis 3: Comparison: Composite; To see the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 1 day after the first treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.002, Regression, Linear — P-value is to test the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 1 day after the first treatment after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = 0.365, 95% CI 2-sided [0.145 to 0.585]

3. Primary Outcome: Change in Urinary Bisphenol A Level (BPA) From Baseline to 14 Days After the First Dental Treatment
Description: BPA was measured, corrected for specific gravity, in ng/mL. We corrected BPA for specific gravity (SG) using the formula: BPA * [(meanSG - 1)/(SG - 1)], where meanSG is the mean of the SG for the samples examined. Urine samples were collected twice pre-treatment and the geometric mean of BPA at each pre-treatment visit was used as the baseline BPA. Change in BPA was computed using BPA at 14 days after the first dental treatment minus BPA at baseline. The first dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically within a few weeks of baseline. Analysis of change in BPA was done using the arithmetic mean.
Time Frame: From Baseline to 14 days after the first dental treatment (The first dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically within a few weeks of baseline.)
Population: Of 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample, 81 subjects who had BPA at 14 days after the first dental treatment were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Composite
Number analyzed (Participants) | 81
ng/mL | -0.50 (4.09)
Statistical Analysis 1: Comparison: Composite; One sample t-test was used to test whether the mean change from baseline was different from 0; Test type: Superiority or Other; p = 0.27, t-test, 2 sided
Statistical Analysis 2: Comparison: Composite; To see the association between composite exposure on all surfaces and change in BPA from baseline to 14 days after the first treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.480, Regression, Linear — P-value is to test the association between composite exposure on all surfaces and change in BPA from baseline to 14 days after the first treatment after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.068, 95% CI 2-sided [-0.258 to 0.123]
Statistical Analysis 3: Comparison: Composite; To see the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 14 days after the first treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.501, Regression, Linear — P-value is to test the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 14 days after the first treatment after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.074, 95% CI 2-sided [-0.293 to 0.145]

4. Primary Outcome: Change in Urinary Bisphenol A Level (BPA) From Baseline to 1 Day After the Second Dental Treatment
Description: BPA was measured, corrected for specific gravity, in ng/mL. We corrected BPA for specific gravity (SG) using the formula: BPA * [(meanSG - 1)/(SG - 1)], where meanSG is the mean of the SG for the samples examined. Urine samples were collected twice pre-treatment and the geometric mean of BPA at each pre-treatment visit was used as the baseline BPA. Change in BPA was computed using BPA at 1 day after the second dental treatment minus BPA at baseline. The second dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically 3-4 weeks after the first dental treatment. Analysis of change in BPA was done using the arithmetic mean.
Time Frame: From Baseline to 1 day after the second dental treatment (The second dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically 3-4 weeks after the first dental treatment.)
Population: Of 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample, 26 subjects who had BPA at 1 day after the second dental treatment were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Composite
Number analyzed (Participants) | 26
ng/mL | -0.59 (3.62)
Statistical Analysis 1: Comparison: Composite; One sample t-test was used to test whether the mean change from baseline was different from 0; Test type: Superiority or Other; p = 0.41, t-test, 2 sided
Statistical Analysis 2: Comparison: Composite; To see the association between composite exposure on all surfaces and change in BPA from baseline to 1 day after the second treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.612, Regression, Linear — P-value is to test the association between composite exposure on all surfaces and change in BPA from baseline to 1 day after the second treatment after adjusting for covariates; [statistical method as in outcome 1, analysis 2]; Slope = -0.082, 95% CI 2-sided [-0.418 to 0.254]
Statistical Analysis 3: Comparison: Composite; To see the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 1 day after the second treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.696, Regression, Linear — P-value is to test the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 1 day after the second treatment after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = 0.078, 95% CI 2-sided [-0.339 to 0.495]

5. Primary Outcome: Change in Urinary Bisphenol A Level (BPA) From Baseline to 14 Days After the Second Dental Treatment
Description: BPA was measured, corrected for specific gravity, in ng/mL. We corrected BPA for specific gravity (SG) using the formula: BPA * [(meanSG - 1)/(SG - 1)], where meanSG is the mean of the SG for the samples examined. Urine samples were collected twice pre-treatment and the geometric mean of BPA at each pre-treatment visit was used as the baseline BPA. Change in BPA was computed using BPA at 14 days after the second dental treatment minus BPA at baseline. The second dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically 3-4 weeks after the first dental treatment. Analysis of change in BPA was done using the arithmetic mean.
Time Frame: From Baseline to 14 days after the second dental treatment (The second dental treatment was scheduled as per treatment needs and the schedules of the dentist and patient. It was typically 3-4 weeks after the first dental treatment.)
Population: Of 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample, 15 subjects who had BPA at 14 days after the second dental treatment were used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Composite
Number analyzed (Participants) | 15
ng/mL | -0.28 (3.55)
Statistical Analysis 1: Comparison: Composite; One sample t-test was used to test whether the mean change from baseline was different from 0; Test type: Superiority or Other; p = 0.76, t-test, 2 sided
Statistical Analysis 2: Comparison: Composite; To see the association between composite exposure on all surfaces and change in BPA from baseline to 14 days after the second treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on all surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.968, Regression, Linear — P-value is to test the association between composite exposure on all surfaces and change in BPA from baseline to 14 days after the second treatment after adjusting for covariates; [statistical method as in outcome 1, analysis 2]; Slope = -0.018, 95% CI 2-sided [-1.061 to 1.025]
Statistical Analysis 3: Comparison: Composite; To see the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 14 days after the second treatment, the linear model was used with the change in BPA outcome. Log-transformed BPA was used for the analysis. Composite exposure on posterior occlusal surfaces was used as the main predictor; Test type: Superiority or Other; p = 0.822, Regression, Linear — P-value is to test the association between composite exposure on posterior occlusal surfaces and change in BPA from baseline to 14 days after the second treatment after adjusting for covariates; Baseline BPA, season, household income, and canned food were used as covariates; Slope = -0.083, 95% CI 2-sided [-0.941 to 0.775]

ADVERSE EVENTS:
Time Frame: It is defined by the time between the first treatment visit and the last study visit (6 months), plus 1 day of observation for Adverse Event.
Description: 91 subjects who had at least one pre-treatment and at least one post-treatment urine sample were used as the total number of subjects at risk. No Adverse Event was reported in this study.
Groups:
- Composite: Restoration of dental caries with dental composite: Dental Resin Restoration (bisphenol A diglycidyl ether methacrylate based composite)
Arm/Group | Composite
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No